CLINICAL TRIAL: NCT01507077
Title: ZGN-440 (Beloranib for Subcutaneous Injection), A Novel Methionine Aminopeptidase 2 Inhibitor for Treatment of Obesity: A Randomized Double-Blind Placebo Controlled Dose Escalation Phase 1b Trial to Evaluate Safety, Pharmacokinetics, Pharmacodynamics and Initial Weight Loss
Brief Title: ZGN-440 (Beloranib for Subcutaneous Injection) for Treatment of Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zafgen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZAF-101
Record Dates: First submitted 2012-01-05; First posted 2012-01-10 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Obesity
Keywords: Obese; Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — CKD732; Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZGN-440 sterile diluent (Placebo Comparator)
  Interventions: Drug: ZGN-440 sterile diluent
- ZGN-440 (Experimental)
  Interventions: Drug: ZGN-440

INTERVENTIONS:
Drug: ZGN-440 — Subjects will receive ZGN-440 twice-weekly over a 4-week treatment period for a total of 8 doses. A range of doses will be evaluated.
  Other Names: Beloranib for subcutaneous injection
  Arms: ZGN-440
Drug: ZGN-440 sterile diluent — Subjects will receive placebo twice-weekly over a 4-week treatment period for a total of 8 doses. A range of doses will be evaluated.
  Arms: ZGN-440 sterile diluent

SUMMARY:
The purpose of this study is to assess the Pharmacokinetics/Pharmacodynamics (PK/PD), safety, and effectiveness of multiple subcutaneous doses of Beloranib (ZGN-440).

DETAILED DESCRIPTION:
This protocol is designed to test the safety and efficacy of a drug called Beloranib (ZGN-440). It is to be tested for its ability to reduce weight in obese female subjects who are of non-childbearing potential. The study will provide information on how much ZGN-440 gets into the blood, how long it stays in the body, and how it affects other biological markers.

ELIGIBILITY:
Inclusion Criteria:

* Obese but otherwise healthy females
* Non-childbearing potential (surgically sterile, post-menopausal, or receiving implanted or injectable contraceptive for at least 3 months)
* BMI ≥ 30 and ≤ 45 kg/m2
* Stable body weight during the past 2 months

Exclusion Criteria:

* Use of weight loss agents in the past month
* History of eating disorder
* History of type 1 or type 2 diabetes mellitus
* Current smokers

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Demonstrate safe doses of ZGN-440 for reduction of body weight in obese female volunteers. | Approximately 4 weeks
  Measures of the safety and tolerability of ZGN-440 include documentation of adverse events and changes (compared to baseline) in vital signs, physical examination, heart rhythm, and laboratory tests.

SECONDARY OUTCOMES:
Incidence, severity and dose-relationship of adverse events as well as changes in physical examinations, ECGs, vital signs and/or laboratory evaluations as a measure of safety and tolerability. | Approximately 4 weeks
Peak plasma concentration of ZGN-440 to assess relationship to weight loss. | Approximately 4 weeks
Elimination half-life of ZGN-440 to assess relationship to weight loss. | Approximately 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: J K Marjason, MD, Principal Investigator — Q-Pharm Clinics, Royal Brisbane and Women's Hospital
Locations (1):
- Q-Pharm Clinics, Royal Brisbane and Women's Hospital, Brisbane, Queensland, Australia